CLINICAL TRIAL: NCT05928390
Title: A Double-blind Randomized Placebo-controlled Dose-finding Phase II Study to Assess the Efficacy and Safety of Pasireotide s.c. in Patients With Post-Bariatric Hypoglycaemia
Brief Title: Pasireotide s.c. in Patients With Post-Bariatric Hypoglycaemia
Acronym: PASIPHY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SOM230-RECAG-CL-0576
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Post-Bariatric Hypoglycemia
Keywords: PBH; Post Bariatric
MeSH Terms: interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pasireotide s.c. 50 mcg (Experimental): Pasireotide 50 mcg s.c. tid
  Interventions: Drug: Pasireotide Diaspartate
- Pasireotide 100 mcg (Experimental): Pasireotide 100 mcg s.c. tid
  Interventions: Drug: Pasireotide Diaspartate
- Pasireotide 200 mcg (Experimental): Pasireotide 200 mcg s.c. tid
  Interventions: Drug: Pasireotide Diaspartate
- Placebo (Placebo Comparator): Placebo s.c. tid
  Interventions: Drug: Pasireotide Diaspartate

INTERVENTIONS:
Drug: Pasireotide Diaspartate — Injectable ampoules
  Other Names: Pasireotide

SUMMARY:
The Total duration of trial participation for each participant with post-bariatric hypoglycemia will be a maximum of 59 weeks, with the following duration of trial periods

* 19 weeks for the Core Phase. It is composed of:

  * a Screening period: a maximum of 3 weeks
  * a Run-in period (no treatment): 4 weeks
  * a Blinded Treatment Phase: 12 weeks
* 36 weeks Extension Phase = an open-label Treatment period
* 4 weeks for the safety follow-up period (without any treatment).

DETAILED DESCRIPTION:
Subjects with post-bariatric hypoglycemia will be screened for participation in this trial. Eligible patients will complete the rest of the Core phase by entering a run-in period of 4 weeks without any treatment.

At the end of the run-in period, participants will be randomized to receive in a blinded manner either pasireotide 50 µg or pasireotide 100 µg or pasireotide 200 µg or Placebo subcutaneously three times a day (prior to each meal).

Participants will blindly self-administer their treatment for a total of 12 weeks when the primary endpoint will be assessed.

All participants completing the core phase will be offered to enter the extension phase. Participants will openly self-administer pasireotide 50 µg or pasireotide 100 µg or pasireotide 200 µg subcutaneously three times a day for a total of 36 weeks of treatment. There will be no more placebo during this extension phase of treatment.

Dose changes/adjustments will be possible only during the extension phase and the decision to change the dose of pasireotide will be left to the investigator's judgment.

All participants will come for a safety visit after discontinuation or completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or- non-pregnant female patients ≥ 18 years of age
2. Patients able to provide and have provided signed written informed consent prior to study participation.
3. Patients capable of self-injecting subcutaneously. Specific training to self-inject the study drug will be provided.
4. Post-bariatric surgery more than 6 months prior to screening
5. Patients with a medically documented diagnosis of PBH and documented glucose measurement (less than 70 mg/dl or 3.9 mmol/L) with symptoms of hypoglycaemia, and resolution following administration of rescue carbohydrates
6. Patients must have ≥ 4 post-prandial hypoglycaemia during the 28-day run-in period (in average ≥1 event over a 7-day week) defined as:

   * Blood glucose less than 54 mg/dL (3.0 mmol/L) as measured by SMBG (level 2) or
   * Level 3 hypoglycaemic event
7. (The previous inclusion criterion number 7 has been deleted).
8. Patients in whom dietary control has not sufficiently controlled symptoms of PBH.
9. Karnofsky Performance Status ≥ 60 (i.e., requires occasional assistance, but is able to care for most of their personal needs)
10. Patients who received other therapies for PBH (such as acarbose, gama guar, pectin, diazoxide) must have stopped all treatments and such treatments are prohibited for a period of at least 2 weeks or 5 half-life times prior to entering the screening period.
11. GLP-1 antagonists and GLP-1 agonists for patients who have been treated with in the past for the indication of PBH, are prohibited for a period of at least 4 weeks before the start of the screening period.
12. SGLT2 inhibitors (glifozins) for patients who have been treated with in the past for the indication of PBH, are prohibited for a period of at least 4 weeks before the start of the screening period.
13. Patients who have been treated with somatostatin receptor analogues in the past, must have an appropriate interval between the last administration of somatostatin receptor analogues treatment and the start of the run-in period as follows:

    * Octreotide s.c. for ≥ 72 hours
    * Octreotide LAR for ≥ 56 days (8 weeks)
    * Lanreotide Autogel for ≥ 98 days (14 weeks)
    * Lanreotide SR ≥ 28 days (4 weeks)
    * Pasireotide s.c. for ≥ 72 hours (3 days)
    * Pasireotide LAR for ≥ 84 days (12 weeks)

Exclusion Criteria :

1. Bariatric patients who have lap band.
2. Patients with a current diagnosis of uncontrolled Diabetes Mellitus. However, diabetic patients in remission, as defined below, are eligible:

   * With an HbA1c at screening less than 6.5%
   * Not taking any medications for hyperglycaemia for at least 3 months prior to screening.
   * Their qualifying Level 3 hypoglycaemia events (see above) must have occurred at least 1 month after the discontinuation of the glucose lowering agent(s).
3. Patients with hypocortisolism, as defined by serum cortisol levels minor of LLN with presence of clinical signs and symptoms of adrenal insufficiency (e.g., weakness, fatigue, anorexia, nausea, vomiting, hypotension, hyponatremia, or hypoglycaemia) as judged by the Investigators
4. (The previous exclusion criterion number 4 has been deleted).
5. (The previous exclusion criterion number 5 has been deleted).
6. Patients who have a known hypersensitivity to somatostatin receptor analogues.
7. Patients currently using medications that may interfere with glucose metabolism within 5 half-lives of drug.
8. Patients with history of or current insulinoma.
9. Patients who have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study such as:

   * Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunodeficiency, including a positive HIV test result (ELISA and Western blot). An HIV test will not be required; however, previous medical history will be reviewed.
   * Non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with this study treatment.
   * Life-threatening autoimmune and ischemic disorders.
   * Inadequate end organ function as defined by:
   * Inadequate bone marrow function:
   * WBC less than 3.0 x 109/L
   * Absolute Neutrophil Count (ANC) less than 1.5 x 109/L
   * Platelets less than100 x 109/L
   * Hgb less than 11 g/dL
   * INR ≥ 1.5
   * eGFR less than 30 mL/min/1.73m2
   * Alkaline phosphatase more than 2.5 x ULN
   * Serum total bilirubin more than1.5 x ULN
   * ALT and AST more than 1.5 x ULN
10. History of liver disease, such as cirrhosis or chronic active hepatitis B andC
11. Presence of Hepatitis B surface antigen (HbsAg) and/ or Presence of Hepatitis C antibody test (anti-HCV). Patients with positive HCV Ab must undergo reflex HCV RNA testing, and patients with HCV RNA positivity will be excluded. Patients with positive HCV Ab and negative HCV RNA are eligible.
12. History of, or current alcohol and/or drug misuse/abuse within the past 12 months. A drug/alcohol test will not be required; however, previous medical history will be reviewed.
13. Patients with symptomatic cholelithiasis and/ or acute or chronic pancreatitis.
14. Patients with abnormal coagulation (PT and PTT elevated by 30% above normal limits).
15. Patients on continuous anticoagulation therapy. Patients who were on anticoagulant therapy must complete a washout period of at least 10 days and have confirmed normal coagulation parameters before study inclusion (patients receiving aspirin once a day are allowed to be enrolled).
16. Patients who are hypothyroid and not on adequate replacement therapy.
17. Patients who have undergone major surgery/surgical therapy for any cause within 1 month before screening. Patients should have recovered from the surgery and be in good clinical condition before entering the study.
18. Patients requiring gastrostomy tube feedings.
19. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study.
20. Clinically significant abnormal laboratory values considered by the Investigator or the medical monitor of the sponsor to be clinically significant or which could have affected the interpretation of the study results.
21. Bradycardia and QT-related exclusion criteria:

    * Patients with long QT syndrome or QTcF more than 450 ms for male and QTcF more than 460 ms for female detected at screening.
    * Patients with uncontrolled or significant cardiac disease, including recent myocardial infarction, unstable angina, congestive heart failure, clinically significant/symptomatic heart rate less than50 bpm, or high-grade AV block, sustained ventricular tachycardia, ventricular fibrillation.
    * History of syncope or family history of idiopathic sudden death.
    * Sustained or clinically significant cardiac arrhythmias.
    * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism, or cardiac failure.
    * Family history of long QT syndrome.
    * Concomitant medications known to prolong the QT interval.
    * Hypokalaemia (Potassium less than or = 3.5 mEq/L).
    * Hypomagnesemia (Magnesium less than 0.7 mmol/L).
22. Participation in any clinical investigation within 4 weeks prior to screening or longer if required by local regulation. (Use of an investigational drug within 1 month prior to screening).
23. Significant acute illness within the two weeks prior to dosing.
24. Female patients who are pregnant, intending to become pregnant or breastfeed during the study. or lactating, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
25. Women of childbearing potential (WOCBP) who are unwilling of using highly effective contraception methods.

    Highly effective contraception methods include:
    * Combined (estrogen and progesterone containing) (oral, intravaginal, transdermal) hormonal contraception associated with inhibition of ovulation.
    * Progesterone-only hormonal (oral, injectable, implantable) contraception associated with inhibition of ovulation.
    * Intrauterine device.
    * Intrauterine hormone-releasing system.
    * Bilateral tubal occlusion.
    * Sexual abstinence defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.
26. Sexually active males unwilling to use a condom during intercourse while taking the drug and for 4 weeks after pasireotide s.c. last dose. A condom is required to be used also by vasectomized men to prevent delivery of the drug via seminal fluid.
27. Potentially unreliable or vulnerable patients (e.g., person kept in detention) and those judged by the Investigator to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the efficacy of pasireotide s.c. on blood glucose concentration during an MMTT in patients with PBH after 12 weeks of treatment. | at baseline and at 12 weeks
  Change in the blood glucose levels, as measured by the peak to nadir glucose AUC during MMTT

SECONDARY OUTCOMES:
KEY SECONDARY_CORE PHASE: Evaluation the change of blood glucose nadir and peak during a mixed meal tolerance test (MMTT) at baseline | at baseline and at 12 weeks
  Change from baseline in the rate of the composite (and individual components) of clinically significant hypoglycaemic events as measured as the frequency of level 2 hypoglycaemic events (glucose level <54 mg/dL or 3.0 mmol/L) measured by SMBG OR the frequency of level 3 hypoglycaemic (requiring external assistance) events/4-weeks at 12 weeks of treatment with pasireotide vs placebo
CORE PHASE: Evaluation of the change of blood glucose nadir and peak during a mixed meal tolerance test (MMTT) at baseline and the MMTT | baseline and 12 weeks
  Change in the nadir and peak of blood glucose levels,
CORE PHASE: Evaluation of the efficacy of pasireotide s.c. on the change from baseline of level 2 hypoglycaemic events during a MMTT in patients with PBH | at 12 weeks
  Change from baseline in the proportion of patients with no level 2 hypoglycaemic events (plasma glucose <54 mg/dL or 3.0 mmol/L) at 60, 90, 105, 120, 135, 150, 165 and 180 min during a 3-hour MMTT
CORE PHASE: Assessessment of the effect of pasireotide s.c. on HRQoL (SF-36 score) | at 12 weeks
  The 36-item Short Form Health Survey (SF-36) is a patient reported outcomes measure that consists of a 36-item self-report inventory. The SF-36 is an accepted metric for benchmarking indications against normative population-based statistics. It assesses health-related limitations in eight dimensions: physical functioning (PF), role limitations due to physical functioning (RP), bodily pain (BP), general health perceptions (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH). Two summary scores, the Physical Component Summary (PCS) and the Mental Component Summary (MCS), can be calculated from the eight-dimension scores (scale scores).
CORE PHASE: Assessessment of the effect of pasireotide s.c. on HRQoL (Dumping Score Questionnaire) | at 12 weeks
  DSQ is a disease specific patient reported outcome (PRO) scale that was developed according to the FDA and EMEA guidelines. The questionnaire utilizes a 5-point Likert scale (0, none; 1, mild; 2, moderate; 3, severe; and 4, very severe) to ask a patient to evaluate the intensity of 10 early dumping symptoms (within 30 minutes (<30 minutes) after food ingestion). In addition, the questionnaire also evaluates 5 late dumping symptoms (more than 1.5 hours (>90 minutes) after food ingestion
CORE PHASE: Assessessment of the effect of pasireotide s.c. on HRQoL (Patient Global Assessment) | at 12 weeks
  It will incorporate a patient global assessment question: "Considering all the way that your disease affects you, rate how you are feeling during the last 7 days compared with your situation before starting the study?" Patients Global Assessment will be measured utilizing a 7-point scale (from 1= a lot worse to 7= a lot better).
CORE PHASE: Assessessment of the effect of pasireotide s.c. on HRQoL (Hypoglycaemia Fear Survey-II) from baseline | at 12 weeks
  The Hypoglycaemia Fear Survey (HFS) originally was developed to measure behaviours and worries related to fear of hypoglycaemia (FOH) in adults with type 1 diabetes. Both the original HFS (HFS-I) and the revised version (HFS-II) are composed of two subscales, the Behaviour (HFS-B) and Worry (HFS-W).
CORE PHASE: Evaluation of the safety profile of pasireotide s.c (AEs) | for 12 weeks
  Incidence of AEs for pasireotide s.c. 50 µg, or 100 µg or 200 µg tid or placebo tid.
EXTENSION PHASE: evaluation of the safety profile of pasireotide s.c. during the whole extension period: (AEs) | for 36 weeks
  Incidence of AEs for pasireotide s.c. 50 µg, or 100 µg or 200 µg tid or placebo tid.
CORE PHASE: Evaluation of the safety profile of pasireotide s.c (Labs) | for 12 weeks
  Incidence of laboratory findings for pasireotide s.c. 50 µg, or 100 µg or 200 µg tid or placebo tid. Changes from baseline in laboratory values and vital signs
EXTENSION PHASE: evaluation of the safety profile of pasireotide s.c. during the whole extension period: (Labs) | for 36 weeks
  Incidence of laboratory findings for pasireotide s.c. 50 µg, or 100 µg or 200 µg tid or placebo tid. Changes from baseline in laboratory values and vital signs
CORE PHASE: Evaluation of the safety profile of pasireotide s.c (ECG) | for 12 weeks
  Incidence of ECG findings for pasireotide s.c. 50 µg, or 100 µg or 200 µg tid or placebo tid. Changes from baseline in ECG readings,
EXTENSION PHASE: evaluation of the safety profile of pasireotide s.c. during the whole extension period: (ECG) | for 36 weeks
  Incidence of ECG findings for pasireotide s.c. 50 µg, or 100 µg or 200 µg tid or placebo tid. Changes from baseline in ECG readings,
CORE PHASE: Evaluation of the safety profile of pasireotide s.c (imaging) | for 12 weeks
  Changes from baseline in gallbladder imaging
EXTENSION PHASE: evaluation of the safety profile of pasireotide s.c. during the whole extension period:(imaging) | for 36 weeks
  Changes from baseline in gallbladder imaging

CONTACTS AND LOCATIONS:
Overall Officials: Arnd H MUELLER, MD, Study Director — Recordati AG
Locations (29):
- United States (10):
  - Stanford University School of Medicine, Endocrinology, 800 Welch Road,, Palo Alto, California
  - Northwestern University - Feinberg School of Medicine - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - NOLA Care, Metairie, Louisiana
  - Velocity Clinical Research - Annapolis, Annapolis, Maryland
  - Joslin Diabetes CenterJoslin Diabetes Center, One Joslin Place, Boston, Massachusetts
  - Mayo Clinic - Rochester, 200 First Street, SW, 55905, Rochester, Minnesota
  - Montefiore Medical Center, 111 E 210th Street,, The Bronx, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at San Antonio, 7703 Floyd Curl Dr,, San Antonio, Texas
  - University of Wisconsin Health W. E. Clinic END, 451 Junction Rd,, Madison, Wisconsin
- Universitaire Ziekenhuizen Leuven, Department of Gastroenterology and Hepatology,Herestraat 49, Leuven, Belgium
- France (3):
  - AP-HP Hopital Europeen Georges Pompidou, 20, rue Leblanc,, Paris
  - HCL Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Rangueil, Attachée de Recherche Clinique, Centre Investigation Clinique, CHU, Cedex 9, France, Toulouse
- Italy (4):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant Orsola, Bologna
  - Azienda Ospedale - Università Padova, Clinica Medica 3, Via Giustiniani, 2,, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, L.go Gemelli 8, Rome
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Passeig Vall d´Hebron 119-129, Spain, Barcelona
  - Hospital Clinic Barcelona, Lipid Clinic End, Nutr. Service Hospital Clinic, C. Villarroel, 170,, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Clinico San Carlos, C/ Prof Martin Lagos s/n, Spain, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (4):
  - North Bristol NHS Trust, Bristol
  - King's College Hospital NHS Foundation Trust, Denmark Hill, SE5 9RS, London
  - Hammersmith Hospital, London
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: Yes